CLINICAL TRIAL: NCT04065438
Title: Treatment of Drug-resistant Adult and Pediatrc Primary Focal Segmental Glomerulosclerosis and Post -Transplant Recurrence Using the LIPOSORBER® LA-15 System
Brief Title: Post Approval Study for Treatment of Drug-resistant Adult and Pediatric Primary FSGS Using the LIPOSORBER® LA-15 System
Acronym: FSGSALLAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaneka Medical America LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMA-FSGS-H170002
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: FSGS; Liposorber
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- LIPOSORBER® LA-15 System (Experimental): All study patients who meet the study eligibility criteria will undergo the extracorporeal treatment using LIPOSORBER® LA-15 System. The participants are to be treated with the system twice weekly for the 3weeks and then once weekly for the following 6 weeks.
  Interventions: Device: LIPOSORBER® LA-15

INTERVENTIONS:
Device: LIPOSORBER® LA-15 — LIPOSORBER® LA-15 is a blood purification therapy; selectively removes apoprotein B-containing lipoproteins such as LDL from circulating blood and rapidly reduces the plasma cholesterol level. It was originally developed for prevention of coronary atherosclerosis progression in patients with serious hyperlipidemia such as familial hypercholesterolemia.
  In the late 1980's, LDL-A was used to improve dyslipidemia in Nephrotic Syndrome, initially to prevent organ damage. LDL-A was found to improve both the dyslipidemic condition and clinical symptoms (proteinuria and hypoproteinemia).

SUMMARY:
This multicenter, prospective, single-arm clinical study will evaluate the probable benefit and safety of the LIPOSORBER® LA-15 System for the treatment of adult patients with nephrotic syndrome associated with primary focal segmental glomerulosclerosis, when the standard treatment options, including corticosteroid and/or calcineurin inhibitors treatments, have been unsuccessful or not well tolerated, and the patient has a GFR ≥ 45 ml/min/1.73m2, or the patient has post-renal transplant recurrence. Treatment for FSGS is considered unsuccessful if the patient is unresponsive to standard therapy (e.g., at least 8 weeks of corticosteroids) and fails to achieve complete or partial remission. A standard treatment is considered not well tolerated if the patient experiences severe side effects without providing an acceptable level of clinical benefit.

DETAILED DESCRIPTION:
This study will enroll up to 35 adult patients at 3-10 clinical sites. The duration of the treatment phase of the study will take approximately 9 weeks for a total of 12 apheresis treatments with the LIPOSORBER® LA-15 System; the treatments will be given twice weekly for 3 weeks followed by once weekly for 6 weeks. Patients will undergo follow-up at 1, 3, 6, 12, and 24 months after the final apheresis treatment.

This study is conducted as a Post Approval Study imposed by Humanitarian Device Exemption (HDE) order to confirm the safety and efficacy of the LIPOSORBER® LA-15 System in the treatment of drug-resistant primary FSGS and post Transplant recurrence.

ELIGIBILITY:
Inclusion Criteria:

A patient is deemed suitable for inclusion in the study if the patient has nephrotic syndrome associated with primary FSGS when:

• Standard treatment options, including corticosteroid and/or calcineurin inhibitors, are unsuccessful or not well tolerated and the patient's glomerular filtration rate (GFR) ≥ 45 ml/min/1.73 m2.

or

• The patient is post renal transplantation.

Exclusion Criteria:

General Exclusion Criteria

1. Patient is greater than 75 years of age at the start of the treatment period or less than 22
2. The patient is unwilling or unable to sign and date the informed consent
3. Pregnant, lactating, or planning to become pregnant prior to completing the study (Note: The safety of the use of LIPOSORBER® in pregnant women has not been studied. There may be unknown risks to an embryo/fetus. Sexually active women of childbearing potential should avoid pregnancy during the use of the LIPOSORBER device and throughout the study duration.)
4. Unable or unwilling to comply with the follow-up schedule
5. Simultaneously participating in another investigational drug or device study
6. Body weight < 15 kg (33.1 lbs)

Medical Exclusion Criteria

1. Currently being administered ACE inhibitors that cannot be withheld for at least 24 hours prior to each apheresis treatment (Note: The time period to withhold ACE inhibitors should be prolonged, if determined by the treating physician, considering each individual's renal function and the biological half-life of the ACE-inhibitor currently in use.)
2. Currently being administered antihypertensive drugs other than ACE inhibitors (e.g., ARBs) that cannot be withheld on the day of apheresis until after the procedure
3. Medical condition or disorder that would limit life expectancy to less than the primary clinical study endpoint or that may cause noncompliance with the study plan or confound the data analysis
4. Hypersensitivity to dextran sulfate, heparin, or ethylene oxide
5. Adequate anticoagulation cannot be achieved due to severe hemophilia, severe hemorrhage diathesis, severe gastrointestinal ulcers, or are recipients of vitamin K antagonist medications
6. Extracorporeal circulation therapy with LIPOSORBER® LA-15 System cannot be tolerated due to severe cardiac insufficiency, acute myocardial infarction, severe cardiac arrhythmia, acute apoplexy, severe uncontrollable hypertension, or severe uncontrollable hypotension Note: Severe uncontrollable hypotension/hypertension indicates the cases with systolic and/or diastolic blood pressure ≤ 5th percentile for age, gender, and height.
7. Cardiac impairments such as uncontrolled arrhythmia, unstable angina, decompensated congestive heart failure, or valvular disease
8. Functional thyroid disease or liver abnormalities
9. Unresolved systemic or local infection that could affect the clinical study outcomes

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and probable benefit of the LIPOSORBER® LA-15 System in relieving nephrotic syndrome associated with primary FSGS at 1 month after the final apheresis treatment. partial remission at 1 month after the final apheresis treatment. | 1 month after the final Apheresis treatment.
  The primary probable benefit endpoint will be assessed by calculating the percent reduction in Up/c values at screening and at 1 month after the final apheresis.

SECONDARY OUTCOMES:
Nephrotic condition at 1, 3, 6, 12, and 24 months after the final apheresis treatment, including the percentage of patients who obtain complete or partial remission at 3, 6, 12, and 24 months. | 1, 3, 6, 12, and 24 months after the final treatment
  Nephrotic condition will be evaluated in following categories, CR (complete remission), PR (partial remission), or NS (nephrotic syndrome).

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Loma Linda University Children's Hospital, Loma Linda, California
  - Loma Linda University Hospital, Loma Linda, California
  - Nemours/Alfred I DuPont Hospital for Children, Wilmington, Delaware
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Weill Cornell Medicine / NewYork-Presbyterian, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Medical University of South Carolina Children's Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Richmond at VCU, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No